CLINICAL TRIAL: NCT01853618
Title: A Pilot Study of Tremelimumab - A Monoclonal Antibody Against CTLA-4 in Combination With Trans-Arterial Catheter Chemoembolization (TACE), Radiofrequency Ablation (RFA), or Cryoablation in Subjects With Hepatocellular Carcinoma (HCC) or Biliary Tract Carcinomas (BTC)
Brief Title: Tremelimumab With Chemoembolization or Ablation for Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 130120; 13-C-0120
Record Dates: First submitted 2013-05-02; First posted 2013-05-15 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Heptocellular Cancer; Biliary Tract Neoplasms; Liver Cancer; Hepatocellular Carcinoma; Biliary Cancer
Keywords: Blocking of Immune Suppression; Monoclonal Antibody; Immunotherapy; Ablative Therapy
MeSH Terms: conditions — Biliary Tract Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — tremelimumab; Radiofrequency Ablation; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Pilot 1/Arm A1-Tremelimumab + RFA or TACE (Experimental): Escalating doses of Tremelimumab + Radiofrequency Ablation (RFA) or Transarterial Catheter Chemoembolization (TACE)
  Interventions: Drug: Tremelimumab; Procedure: RFA; Procedure: TACE
- 2/Arm A2 - Tremelimumab + RFA or TACE (Experimental): Tremelimumab + Radiofrequency Ablation (RFA) or Transarterial Catheter Chemoembolization (TACE)
  Interventions: Drug: Tremelimumab; Procedure: RFA; Procedure: TACE
- 3/Arm B - Tremelimumab + TACE (Experimental): Tremelimumab + Transarterial Catheter Chemoembolization (TACE)
  Interventions: Drug: Tremelimumab; Procedure: TACE
- 4/Arm C (never opened) (Experimental): Tremelimumab + Radiofrequency Ablation (RFA) or Transarterial Catheter Chemoembolization (TACE)
  Interventions: Drug: Tremelimumab; Procedure: TACE; Procedure: Cryoablation
- 5/Arm D - Tremelimumab + Cryoablation (Experimental): Tremelimumab + Cryoablation
  Interventions: Drug: Tremelimumab; Procedure: Cryoablation
- 6/Arm E - Tremelimumab + RFA (Experimental): Tremelimumab + Radiofrequency Ablation (RFA)
  Interventions: Drug: Tremelimumab; Procedure: RFA

INTERVENTIONS:
Drug: Tremelimumab — 3.5 mg/kg or 10 mg /kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  Other Names: Ticilimumab
Procedure: RFA — Performed on Day 36
  Other Names: Radiofrequency Ablation
  Arms: 2/Arm A2 - Tremelimumab + RFA or TACE; 6/Arm E - Tremelimumab + RFA; Pilot 1/Arm A1-Tremelimumab + RFA or TACE
Procedure: TACE — Performed on Day 36 and may be repeated (as per standard of care) on months 3, 7, and 13, and every (q)6 months thereafter (if indicated)
  Other Names: Transarterial Catheter Chemoembolization
  Arms: 2/Arm A2 - Tremelimumab + RFA or TACE; 3/Arm B - Tremelimumab + TACE; 4/Arm C (never opened); Pilot 1/Arm A1-Tremelimumab + RFA or TACE
Procedure: Cryoablation — Performed on Day 36
  Arms: 4/Arm C (never opened); 5/Arm D - Tremelimumab + Cryoablation

SUMMARY:
Background:

- Tremelimumab is a cancer treatment drug that helps the immune system recognize and destroy cancer cells. Researchers want to see if it can be used to treat advanced liver cancer. The drug will be given with one of two types of treatment for liver cancer. The first type, transarterial catheter chemoembolization (TACE), injects chemotherapy drugs into the tumor through the main blood vessel that is feeding it. That blood vessel is then closed off to help keep the drugs in the tumor longer. The second type, radiofrequency ablation (RFA), uses a heated probe to destroy the tumor tissue. Researchers want to study how safe and effective these treatments are with the study drug.

Objectives:

- To test the safety and effectiveness of Tremelimumab with TACE or RFA for advanced liver cancer.

Eligibility:

- Individuals at least 18 years of age who have advanced liver cancer that has not responded to other treatments.

DETAILED DESCRIPTION:
Background:

Worldwide, hepatocellular carcinoma (HCC) is the fifth most common malignancy with a median survival of 6-9 months. For patients with advanced disease sorafenib is the only approved drug and this has limited benefit.

Tremelimumab is a monoclonal antibody against cytotoxic T-lymphocyte-associated protein 4 (CTLA4). Anti-CTLA4 therapy has been shown to enhance anti-tumor immunity by blocking tumor-induced immune suppression of cytotoxic T cells.

Various tumor ablative procedures and techniques have been shown to result in immunogenic cell death and induction of a peripheral immune response. Both transarterial catheter chemoembolization (TACE) and radiofrequency ablation (RFA) have been shown to do this, as well as cryoablation and external beam radiation.

The underlying hypothesis of this study is that the effect of anti-CTLA4 treatment can be enhanced by TACE or RFA in patients with advanced hepatocellular carcinoma. We will also evaluate this in the context of cryoablation and radiation in hepatocellular carcinoma (HCC) and RFA in cholangiocarcinoma.

Objective:

To assess the safety and feasibility of combining Tremelimumab with trans-arterial catheter chemoembolization (TACE) radiofrequency ablation (RFA), or cryoablation in patients with advanced HCC.

Eligibility:

Histologically or cytologically confirmed diagnosis of HCC.

Childs-Pugh A/B7 cirrhosis only is allowed. If patient does not have cirrhosis, this limitation does not apply.

Barcelona Clinic Liver Cancer (BCLC) Stage B and C patients.

Patients must have disease that is not amenable to potentially curative resection, radiofrequency ablation, or liver transplantation.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have histopathological confirmation of hepatocellular carcinoma (HCC) or (Cohort E only) biliary tract carcinoma (BTC) by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study OR histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of HCC (or biliary tract carcinoma in Cohort E). Fibrolammelar variant is also allowed. For cohort E, the term BTC includes intraor extrahepatic cholangiocarcinoma, gallbladder cancer or ampullary cancer, as long as there is an intrahepatic component amenable to radiofrequency ablation (RFA).
2. Patients must have disease that is not amenable to potentially curative resection, transplantation or ablation. For Cohorts A, C and D patients must have progressed on, been intolerant to, or refused prior sorafenib therapy. Cohort E patients must have received at least one line of chemotherapy for BTC.
3. Disease must be technically amenable to transhepatic arterial chemoembolization (TACE), radiofrequency ablation (RFA) or cryoablation. Each case will be discussed at gastrointestinal (GI) tumor board with interventional radiology. Patients must have evaluable disease.
4. If liver cirrhosis is present, patient must have a Child-Pugh A/B7 classification.
5. Age greater than or equal to 18 years
6. Life expectancy of greater than 3 months.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
8. Patients must have normal organ and marrow function as defined below:

   * leukocytes greater than or equal to 3,000/mcL
   * absolute neutrophil count greater than or equal to 1,000/mcL
   * platelets greater than or equal to 60,000/mcL
   * total bilirubin, If cirrhosis present: Part of Child Pugh requirement. If no cirrhosis: Bili should be less than or equal to 2 times upper limit of normal (ULN)
   * Serum albumin, If cirrhosis present: Part of Child Pugh requirement. If no cirrhosis: albumin should be greater than or equal to 2.5g/dl
   * Patients are eligible with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) up to 5 times ULN.
   * creatinine, less than 1.5 times institution upper limit of normal OR
   * creatinine clearance greater than or equal to 45 mL/min/1.73 m(2), as calculated below, for patients with creatinine levels above institutional normal
9. Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.
10. Patients must not have other invasive malignancies within the past 5 years (with the exception of non-melanoma skin cancers, non-invasive bladder cancer or localized prostate cancer for whom systemic therapy is not required).
11. Patient must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients who have had standard of care chemotherapy, large field radiotherapy, or major surgery must wait 2 weeks prior to entering the study. For recent experimental therapies a 28 day period of time must elapse before treatment.
2. Patients who have undergone prior liver transplantation are ineligible.
3. Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations that would limit compliance with study requirements.
5. History of chronic autoimmune disease (e.g., Addison's disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, rheumatoid arthritis, hypophysitis, etc.) with symptomatic disease within the 3 years before randomization. Note: Active vitiligo or a history of vitiligo will not be a basis for exclusion.
6. Dementia or significantly altered mental status that would prohibit the understanding or rendering of Information and Consent and compliance with the requirements of the protocol.
7. Diverticulitis (either active or history of) within the past 2 years. Note that diverticulosis is permitted.
8. Active or history of inflammatory bowel disease (colitis, Crohn's), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegener's granulomatosis.
9. Currently receiving immunosuppressive doses of steroids or other immunosuppressive medications (inhaled and topical steroids are permitted)
10. History of sarcoidosis syndrome
11. Patients should not be vaccinated with live attenuated vaccines within 1 month of starting Tremelimumab treatment.

12 Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)

13. HIV-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and Tremelimumab. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that Tremelimumab may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events.

14. History of hypersensitivity reaction to human or mouse antibody products.

15. Pregnancy and breast feeding are exclusion factors. The effects of Tremelimumab on the developing human fetus are unknown. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

16. Patients with unhealed surgical wounds for more than 30 days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-05-02 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Result] Xie C, Duffy AG, Mabry-Hrones D, Wood B, Levy E, Krishnasamy V, Khan J, Wei JS, Agdashian D, Tyagi M, Gangalapudi V, Fioravanti S, Walker M, Anderson V, Venzon D, Figg WD, Sandhu M, Kleiner DE, Morelli MP, Floudas CS, Brar G, Steinberg SM, Korangy F, Greten TF. Tremelimumab in Combination With Microwave Ablation in Patients With Refractory Biliary Tract Cancer. Hepatology. 2019 May;69(5):2048-2060. doi: 10.1002/hep.30482. Epub 2019 Mar 10. PMID 30578687
- [Result] Agdashian D, ElGindi M, Xie C, Sandhu M, Pratt D, Kleiner DE, Figg WD, Rytlewski JA, Sanders C, Yusko EC, Wood B, Venzon D, Brar G, Duffy AG, Greten TF, Korangy F. The effect of anti-CTLA4 treatment on peripheral and intra-tumoral T cells in patients with hepatocellular carcinoma. Cancer Immunol Immunother. 2019 Apr;68(4):599-608. doi: 10.1007/s00262-019-02299-8. Epub 2019 Jan 28. PMID 30688989
- [Result] Duffy AG, Ulahannan SV, Makorova-Rusher O, Rahma O, Wedemeyer H, Pratt D, Davis JL, Hughes MS, Heller T, ElGindi M, Uppala A, Korangy F, Kleiner DE, Figg WD, Venzon D, Steinberg SM, Venkatesan AM, Krishnasamy V, Abi-Jaoudeh N, Levy E, Wood BJ, Greten TF. Tremelimumab in combination with ablation in patients with advanced hepatocellular carcinoma. J Hepatol. 2017 Mar;66(3):545-551. doi: 10.1016/j.jhep.2016.10.029. Epub 2016 Nov 2. PMID 27816492
- [Result] Greten TF, Sangro B. Targets for immunotherapy of liver cancer. J Hepatol. 2017 Sep 18:S0168-8278(17)32287-0. doi: 10.1016/j.jhep.2017.09.007. Online ahead of print. PMID 28923358
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0120.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4/Arm C never opened, thus no participants were enrolled in this group.
Groups:
- Pilot 1/Arm A1-Tremelimumab + RFA or TACE: Escalating doses of Tremelimumab + Radiofrequency Ablation (RFA) or Transarterial Catheter Chemoembolization (TACE)
  Tremelimumab: 3.5 mg/kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  RFA: Performed on Day 36
  TACE: Performed on Day 36 and may be repeated (as per standard of care) on months 3, 7, and 13, and every (q)6 months thereafter (if indicated)
- 2/Arm A2 - Tremelimumab + RFA or TACE: Tremelimumab + Radiofrequency Ablation (RFA) or Transarterial Catheter Chemoembolization (TACE)
  Tremelimumab: 10 mg /kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  RFA: Performed on Day 36
  TACE: Performed on Day 36 and may be repeated (as per standard of care) on months 3, 7, and 13, and every (q)6 months thereafter (if indicated)
- 3/Arm B - Tremelimumab + TACE: Tremelimumab + Transarterial Catheter Chemoembolization (TACE)
  Tremelimumab: 10 mg /kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  TACE: Performed on Day 36 and may be repeated (as per standard of care) on months 3, 7, and 13, and every (q)6 months thereafter (if indicated)
- 5/Arm D - Tremelimumab + Cryoablation: Tremelimumab + Cryoablation
  Tremelimumab: 10 mg /kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  Cryoablation: Performed on Day 36
- 6/Arm E - Tremelimumab + RFA: Tremelimumab + Radiofrequency Ablation (RFA)
  Tremelimumab: 10 mg /kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  RFA: Performed on Day 36
Period: Overall Study
Arm/Group | Pilot 1/Arm A1-Tremelimumab + RFA or TACE | 2/Arm A2 - Tremelimumab + RFA or TACE | 3/Arm B - Tremelimumab + TACE | 5/Arm D - Tremelimumab + Cryoablation | 6/Arm E - Tremelimumab + RFA
Started | 8 | 12 | 12 | 9 | 20
Completed | 6 | 10 | 10 | 8 | 17
Not Completed | 2 | 2 | 2 | 1 | 3
Not completed — Bile duct stent blockage/progressive dis | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 1 | 1 | 1 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot 1/Arm A1-Tremelimumab + RFA or TACE | 2/Arm A2 - Tremelimumab + RFA or TACE | 3/Arm B - Tremelimumab + TACE | 5/Arm D - Tremelimumab + Cryoablation | 6/Arm E - Tremelimumab + RFA | Total
Number analyzed (Participants) | 8 | 12 | 12 | 9 | 20 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 12 | 9 | 3 | 18 | 48
  >=65 years | 2 | 0 | 3 | 6 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.53 (15.27) | 64.02 (10.4) | 55.68 (10.17) | 64.12 (11.73) | 55.79 (8.89) | 59.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 0 | 10 | 14
  Male | 6 | 12 | 10 | 9 | 10 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 7 | 12 | 11 | 9 | 20 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 7 | 5 | 0 | 14
  White | 2 | 12 | 4 | 3 | 20 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 12 | 9 | 20 | 61
Previous Therapy [Count of Participants; unit: Participants] — Transarterial catheter chemoembolization (TACE)
  Participants
    Any surgical resection | 3 | 1 | 2 | 3 | 10 | 19
    Any TACE | 2 | 5 | 0 | 2 | 0 | 9
    Any chemotherapy | 8 | 12 | 11 | 9 | 20 | 60
    Any radiation therapy | 3 | 2 | 0 | 0 | 4 | 9
    Misc. therapy - Y90 | 1 | 2 | 0 | 0 | 0 | 3
    Misc. therapy - Hyperthermia | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-Serious Adverse Events Regardless of Attribution
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 44 months and 5 days for 1/Arm A1; 49 months and 26 days for 2/Arm A2; 1 month and 26 days for 3/Arm B; 30 months and 20 days for 5/Arm D; and 34 months and 25 days for 6/Arm E.
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot 1/Arm A1-Tremelimumab + RFA or TACE | 2/Arm A2 - Tremelimumab + RFA or TACE | 3/Arm B - Tremelimumab + TACE | 5/Arm D - Tremelimumab + Cryoablation | 6/Arm E - Tremelimumab + RFA
Number analyzed (Participants) | 8 | 12 | 12 | 9 | 20
Participants | 8 | 12 | 12 | 9 | 20

2. Secondary Outcome: Number of Participants With Best Response
Description: Best response was assessed by the combined Response Evaluation Criteria in Solid Tumors (RECIST and the Modified Immune-Related Response Criteria (irRC). Complete Response (CR) is disappearance of all target lesions. Any patjhological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if it is the smallest on study). The appearance of one or more lesions is also considered progressions.
Time Frame: Start of study, baseline target lesions until disease progression occurs with 20% increase of target lesions or appearance of new lesions, up to 13.1 months
Measure: Count of Participants; unit: Participants
Groups:
- 6/Arm E - Tremelimumab + RFA: Tremelimumab + Radiofrequency Ablation (RFA)
  Tremelimumab:10 mg /kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  RFA: Performed on Day 36
Arm/Group | Pilot 1/Arm A1-Tremelimumab + RFA or TACE | 2/Arm A2 - Tremelimumab + RFA or TACE | 3/Arm B - Tremelimumab + TACE | 5/Arm D - Tremelimumab + Cryoablation | 6/Arm E - Tremelimumab + RFA
Number analyzed (Participants) | 8 | 12 | 12 | 9 | 20
Participants
  Complete Response | 0 | 0 | 1 | 0 | 0
  Partial Response | 1 | 2 | 2 | 2 | 2
  Stable Disease | 3 | 5 | 4 | 3 | 5
  Progressive Disease | 1 | 3 | 4 | 3 | 11
  Not Evaluable | 3 | 2 | 1 | 1 | 2

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the amount of time a subject survives without disease progression after treatment. Progression is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if it is the smallest on study). The appearance of one or more lesions is also considered progressions.
Time Frame: Progression free survival is time patients were off treatment until death. For all cohorts progression free survival ranged from 3.4 months to 8.6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pilot 1/Arm A1-Tremelimumab + RFA or TACE | 2/Arm A2 - Tremelimumab + RFA or TACE | 3/Arm B - Tremelimumab + TACE | 5/Arm D - Tremelimumab + Cryoablation | 6/Arm E - Tremelimumab + RFA
Number analyzed (Participants) | 8 | 12 | 12 | 9 | 20
Months | 6.4 [0.8 to 12] | 7.5 [5.6 to 9.3] | 7.7 [5.8 to 9.5] | 8.6 [2.8 to 15.5] | 3.4 [2.5 to 5.2]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the amount of time a subject survives after therapy.
Time Frame: From the time of initial treatment consent until date of death for each patient. Overall survival ranged from 6 months to 13.1 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pilot 1/Arm A1-Tremelimumab + RFA or TACE | 2/Arm A2 - Tremelimumab + RFA or TACE | 3/Arm B - Tremelimumab + TACE | 5/Arm D - Tremelimumab + Cryoablation | 6/Arm E - Tremelimumab + RFA
Number analyzed (Participants) | 8 | 12 | 12 | 9 | 20
Months | 10.5 [5.2 to 15.7] | 8.4 [6.5 to 10.3] | 13.1 [11.3 to 15] | 13.1 [6.3 to 19.9] | 6 [3.8 to 8.8]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 44 months and 5 days for 1/Arm A1-Tremelimumab + RFA or TACE; 49 months and 26 days for 2/Arm A2-MTD of Tremelimumab + RFA or TACE; 1 month and 26 days for 3/Arm B-MTD of Tremelimumab + TACE; 30 months and 20 days for 5/Arm D-MTD of Tremelimumab + Cryoablation; and 34 months and 25 days for 6/Arm E-MTD of Tremelimumab + RFA.
Description: All deaths in the mortality module are attributable to progressive disease (all deaths that occurred are reported).
Groups:
- 2/Arm A2 -Tremelimumab + RFA or TACE: Tremelimumab + Radiofrequency Ablation (RFA) or Transarterial Catheter Chemoembolization (TACE)
  Tremelimumab: 10 mg /kg intravenous (IV) every 4 weeks times 6 doses and then every 12 weeks for 2 years
  RFA: Performed on Day 36
  TACE: Performed on Day 36 and may be repeated (as per standard of care) on months 3, 7, and 13, and every (q)6 months thereafter (if indicated)
Arm/Group | Pilot 1/Arm A1-Tremelimumab + RFA or TACE | 2/Arm A2 -Tremelimumab + RFA or TACE | 3/Arm B - Tremelimumab + TACE | 5/Arm D - Tremelimumab + Cryoablation | 6/Arm E - Tremelimumab + RFA
All-Cause Mortality (participants affected / at risk) | 8/8 | 1/12 | 8/12 | 6/9 | 17/20
Serious Adverse Events (participants affected / at risk) | 5/8 | 1/12 | 7/12 | 3/9 | 7/20
Other Adverse Events (participants affected / at risk) | 8/8 | 12/12 | 12/12 | 9/9 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot 1/Arm A1-Tremelimumab + RFA or TACE (N=8) | 2/Arm A2 -Tremelimumab + RFA or TACE (N=12) | 3/Arm B - Tremelimumab + TACE (N=12) | 5/Arm D - Tremelimumab + Cryoablation (N=9) | 6/Arm E - Tremelimumab + RFA (N=20)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, HCC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Gastrointestinal disorders - Other, Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, C. Diff. (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Blackout (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, C. Diff. (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot 1/Arm A1-Tremelimumab + RFA or TACE (N=8) | 2/Arm A2 -Tremelimumab + RFA or TACE (N=12) | 3/Arm B - Tremelimumab + TACE (N=12) | 5/Arm D - Tremelimumab + Cryoablation (N=9) | 6/Arm E - Tremelimumab + RFA (N=20)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (19) | 4 (8) | 12 (21)
Activated partial thromboplastin time prolonged (Investigations) | 4 (15) | 10 (11) | 9 (20) | 4 (6) | 14 (26)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (33) | 1 (5) | 10 (33) | 7 (16) | 8 (16)
Alkaline phosphatase increased (Investigations) | 7 (27) | 1 (2) | 10 (43) | 5 (12) | 13 (25)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 8 (31) | 12 (17) | 11 (68) | 9 (31) | 20 (73)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 6 (11) | 5 (9) | 2 (2) | 8 (11)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (7) | 1 (2) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 8 (46) | 1 (1) | 10 (55) | 8 (25) | 13 (39)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (3) | 1 (1) | 4 (6)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Blood bilirubin increased (Investigations) | 6 (24) | 1 (2) | 8 (35) | 4 (14) | 7 (21)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (9) | 8 (12) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 5 (8) | 1 (1) | 5 (5)
Creatinine increased (Investigations) | 3 (3) | 1 (7) | 6 (20) | 4 (17) | 7 (15)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (7) | 4 (4) | 2 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 6 (12) | 2 (4) | 9 (16)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (5) | 5 (5) | 3 (6)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (5) | 6 (12) | 8 (13) | 2 (5) | 12 (18)
Fever (General disorders) | 3 (3) | 1 (2) | 7 (9) | 1 (1) | 11 (20)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Dry throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (27) | 10 (44) | 11 (74) | 7 (29) | 16 (60)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 3 (5) | 3 (5) | 6 (10)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 5 (14) | 6 (16) | 8 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (7) | 2 (2) | 3 (17) | 2 (9) | 7 (11)
Hyponatremia (Metabolism and nutrition disorders) | 8 (19) | 12 (40) | 12 (44) | 6 (25) | 12 (31)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 9 (38) | 5 (7) | 8 (21)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, Oral thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 7 (7) | 1 (1) | 3 (4)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, HCC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (5) | 0 (0) | 3 (3) | 8 (14)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (11) | 0 (0) | 5 (8) | 1 (1) | 9 (11)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 6 (27) | 3 (15) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, mouth ulcers (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (8) | 2 (2) | 4 (5)
Weight loss (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 4 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (5) | 1 (4) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, gastrointestinal disorders - Other, cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (4) | 1 (2) | 1 (1)
Hoarseness: voice changes (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypersomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin peeling - bil. Hands (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, atrial fib with bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 5 (8) | 2 (4) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Infections and infestations - Other, Infection - E.coli (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (18) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, blisters on abdominal area (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, various scabs (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delayed orgasm (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (3) | 2 (5) | 3 (3) | 6 (7)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, neuro-gait abnormalities (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (5) | 2 (2) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1) | 5 (7) | 3 (6) | 8 (32)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (13)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Infections and infestations - Other, C. Diff infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Infections and infestations - Other, Infection-GI other, liver infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (32) | 6 (31) | 11 (68) | 7 (23) | 17 (63)
Lymphocyte count increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 6 (16) | 8 (15) | 2 (3) | 4 (6)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 2 (4) | 1 (14) | 3 (7)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 5 (11) | 4 (17) | 8 (34) | 6 (10) | 13 (26)
Platelet count decreased (Investigations) | 5 (25) | 3 (12) | 5 (22) | 5 (15) | 9 (22)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — - Other, skin and subcutaneous tissue disorders - Other: skin lesions
Skin and subcutaneous tissue disorders - Other, lymph node swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT01853618/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT01853618/ICF_001.pdf